CLINICAL TRIAL: NCT01214070
Title: Functional Vision Consequences of Rehabilitation for TBI Vision Loss
Brief Title: Functional Vision in TBI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative Closure
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C6687-R
Record Dates: First submitted 2010-09-14; First posted 2010-10-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Brain Injuries; Visually Impaired Persons
Keywords: Visual Perception; Vision, Ocular; Neuronal Plasticity
MeSH Terms: conditions — Brain Injuries | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm 1 (Active Comparator): Group 1 - Combination Treatment
  Interventions: Other: Vision Restoration Therapy; Behavioral: NVT Eye Scanning Therapy
- Arm 2 (Active Comparator): Group 2 - Combination Treatment
  Interventions: Behavioral: Eccentric Viewing Training
- Arm 3 (Active Comparator): Group 3 - Combination Treatment
  Interventions: Other: Vision Restoration Therapy; Behavioral: NVT Eye Scanning Therapy
- Arm 4 (Active Comparator): Group 4 - Combination Treatment
  Interventions: Behavioral: Eccentric Viewing Training
- Arm 5 (Active Comparator): Group 5 - Monotherapy Treatment
  Interventions: Other: Vision Restoration Therapy; Behavioral: Sham
- Arm 6 (Active Comparator): Group 6 - Monotherapy Treatment
  Interventions: Behavioral: Eccentric Viewing Training; Behavioral: Sham
- Arm 7 (Active Comparator): Group 7 - Monotherapy Treatment
  Interventions: Behavioral: NVT Eye Scanning Therapy; Behavioral: Sham

INTERVENTIONS:
Other: Vision Restoration Therapy — Therapy that enhances the neuronal plasticity of the visual system
  Arms: Arm 1; Arm 3; Arm 5
Behavioral: NVT Eye Scanning Therapy — Therapy that trains eye and head scanning into the blind hemianoptic visual field
  Arms: Arm 1; Arm 3; Arm 7
Behavioral: Eccentric Viewing Training — Therapy that trains the person to compensate for visual field loss by learning to move the visual field loss to the position that is least likely to impact the current visual task
  Arms: Arm 2; Arm 4; Arm 6
Behavioral: Sham — Therapy that encourages subjects to do daily visual tasks at home while having no training or intended intervention benefit
  Arms: Arm 5; Arm 6; Arm 7

SUMMARY:
The objective of this study is to test functional vision outcome measures that reflect the loss in everyday life tasks that require vision and that are sensitive to changes after a course of vision rehabilitation in Veterans/participants with TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) can cause vision loss because of diffuse or focal neuronal injury. Vision can be compromised because of local injury to one or both optic nerves, diffuse brain injury, and/or limitation in eye movements because of dysfunction of cranial nerves. These typical injuries may compromise any of the neural pathways that subserve afferent or efferent visual function. Self-reports of vision loss include diplopia, visual field loss, light sensitivity, reading problems and contrast sensitivity (color and luminance) loss. This project will pursue the following aims: 1) Identify the relationship between functional vision loss in everyday vision tasks (reading, visual search, way finding) and the characteristics of potential visual impairment (visual acuity, contrast sensitivity, visual fields, stereoacuity, eye movement disorders) associated with TBI; and 2) Determine the ability of the vision rehabilitation interventions (both monotherapy and combination therapy) to improve functional vision outcome measures that reflect everyday visual tasks. The vision rehabilitation interventions incorporated into this study will be Vision Restoration Therapy, NVT Eye Scanning Therapy, and standard Eccentric Viewing Training. These therapies are rehabilitative interventions prescribed for Veterans in Polytrauma Rehabilitation Centers, Blind Rehabilitation Centers, and advocated for VA Medical Center TBI clinics.

ELIGIBILITY:
Inclusion Criteria:

* TBI (any form)
* Hemianopic Visual Field Loss
* Stable fixation
* 1.0 logMAR or better Reading Acuity
* 20 words per minute or better reading rate

Exclusion Criteria:

* Visual Neglect
* medical conditions that prevent sitting for 30 minutes or following instructions

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-06-01 (Actual); Primary Completion 2013-11-21 (Actual); Study Completion 2013-11-21 (Actual)

PRIMARY OUTCOMES:
Dynamic Visual Field | Baseline

SECONDARY OUTCOMES:
Dynamic Visual Field | After First Therapy / Before Second Therapy (Average time is 4.5 months)
Dynamic Visual Field | After Second Therapy (Average Time is 9 months)
Reading Rate and Accuracy | Baseline
Reading Rate | After First Therapy / Before Second Therapy (average time is 4.5 months)
Reading Rate and Accuracy | After Second Therapy (average time is 9 months)
Visual Search Accuracy and Timing | Baseline
Visual Search Accuracy and Timing | After First Therapy / Before Second Therapy (average time is 4.5 months)
Visual Search Accuracy and Timing | After Second Therapy (average time is 9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Schuchard, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States